CLINICAL TRIAL: NCT07159945
Title: Controlling Nutritional Status as a Superior Predictor of Fixation Failure in Intertrochanteric Fractures: Development and Validation of a Multicentre Nomogram
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Fang, Deputy chief physician, First Affiliated Hospital of Fujian Medical University
Other Study IDs: MTCA,ECFAH Of FMU [2015]084 -2
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Intertrochanteric Fractures; Internal Fixation Failure; CONUT Score; Nomogram Model; Nutritional Status
Keywords: Intertrochanteric Fractures; Internal fixation failure; CONUT score; Nomogram model; Nutritional Status
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FIF-ITF group
- Control group

SUMMARY:
A multicentre retrospective cohort study was conducted within the Department of Orthopaedics at the First Affiliated Hospital of Fujian Medical University. This study reviewed 1,296 patients who underwent internal fixation treatment with ITF at the institution between 2020 and 2024. This study employed three distinct nutritional assessment tools for preoperative nutritional evaluation: CONUT, PNI, and NPS. By comparing the prevalence of malnutrition across these three scales and their relationship with FIF-ITF, an optimal predictive model combining INST with clinical factors was established.

DETAILED DESCRIPTION:
A multicentre retrospective cohort study was conducted within the Department of Orthopaedics at the First Affiliated Hospital of Fujian Medical University. This study reviewed 1,296 patients who underwent internal fixation treatment with ITF at the institution between 2020 and 2024. Detailed documentation of patient information, including age, gender, affected side, bone mineral density (BMD), age-adjusted Charlson Comorbidity Index (aCCI), fracture type, internal fixation method, haematological parameters, implant-related complications (INSTs), and reasons for failure. This study employed three distinct nutritional assessment tools for preoperative nutritional evaluation: CONUT, PNI, and NPS. By comparing the prevalence of malnutrition across these three scales and their relationship with FIF-ITF, an optimal predictive model combining INST with clinical factors was established.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of ITF on the basis of medical history, symptoms, imaging data, etc.; 2. Treatment by internal fixation surgery; 3. Normal cognitive function; and 4. Informed consent obtained from the patient or family.

Exclusion Criteria:

* 1. Significant missing data: In accordance with the Transparent Reporting of a Multivariate Prediction Model for Individual Prognosis or Diagnosis (TRIPOD) statement, only cases with complete key variables (missing rate <5%) were included; 2. Severe preoperative systemic comorbidities (e.g., decompensated liver/renal failure, active pneumonia, malignancy, and cachexia) and/or a history of mental illness; and 3. Missing postoperative follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to inclusion criteria, 1,296 patients undergoing internal fixation for intertrochanteric fractures at the aforementioned medical institutions between 2020 and 2024 were selected. All patients completed at least one year of follow-up. Follow-up comprised comprehensive orthopaedic examinations and serological tests, supplemented by repeat imaging where necessary to assess local fracture/internal fixation status.
Sampling Method: Non-Probability Sample
Enrollment: 1296 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The CONUT score | Before surgery
The PNI score | Before surgery
The NPS score | Before surgery

SECONDARY OUTCOMES:
serum albumin | Before surgery
total cholesterol | Before surgery
lymphocyte count | Before surgery
fracture type | Before surgery
age | Before surgery
osteoporosis | Before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Liu Zhang, MD, Study Director — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China